CLINICAL TRIAL: NCT01795339
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Two-Part, Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Effect on Biomarkers of AZD3293 in Plasma and Cerebrospinal Fluid in Healthy Male and Non-Fertile Female Elderly Volunteers and in Mild-to-Moderate Alzheimer Disease Patients
Brief Title: A Two-part Multiple Dose Study to Assess the Safety and Effects of AZD3293 in Healthy Elderly and Alzheimer's Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D5010C00002
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Healthy Elderly Volunteers; Mild-to-moderate Alzheimer's Disease Patients
Keywords: AZD3293; Healthy volunteers; Elderly volunteers; Alzheimer's Disease patients; AD patients; Phase 1; Multiple Ascending Dose Study
MeSH Terms: interventions — lanabecestat

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- AZD3293 (Experimental): Part 1: Up to 6 sequential cohorts of healthy elderly subjects are planned, with multiple ascending doses, starting with 5 mg (subject to confirmation by the Safety Review Committee) Part 2: Up to 16 mild-to-moderate AD patients administered one to up to 3 dosage levels of AZD3293
  Interventions: Drug: AZD3293
- Placebo (Placebo Comparator): Part 1: Placebo given (2 subjects in each cohort) Part 2: Placebo given (up to 4 subjects)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD3293 — Oral solution
  Arms: AZD3293
Drug: Placebo — Oral solution
  Arms: Placebo

SUMMARY:
This is a two-part multiple dose study in healthy male and female (of non-child bearing potential) elderly volunteers, and in Alzheimer's disease patients, to assess the safety, effects on the body, and blood, CSF, and urine drug levels of AZD3293. AZD3293 is being developed for the treatment of Alzheimer's Disease

DETAILED DESCRIPTION:
A Phase I, Randomized, Double-Blind, Placebo-Controlled, Two-Part, Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Effect on Biomarkers of AZD3293 in Plasma and Cerebrospinal Fluid in Healthy Male and Non-Fertile Female Elderly Volunteers and in Mild-to-Moderate Alzheimer Disease Patients

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Healthy elderly male and female (of non-childbearing potential) subjects.
* Part 2: Male and non-fertile female AD patients.
* Body mass index (BMI) between 19 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg.
* Part 2: Clinical diagnosis of probable AD according to the NINCDS-ADRDA criteria.
* Part 2: Manifestation of AD symptoms at least 6 months before randomization.

Exclusion Criteria:

* Part 1: History or presence of psychiatric disease/condition, GI, renal, hepatic, cardiovascular, psychiatric, or retinal diseases or disorders.
* Part 2: Significant disease affecting the CNS other than Alzheimer's disease, including but not limited to other dementias, other significant neurological or major psychiatric disease.
* History of use of antipsychotic drugs , or chronic use of antidepressant or anxiolytic drugs.
* Frequent use (more than 2 days per week during the last 12 weeks) of tobacco or other nicotine products.
* History of neurological disease, including seizures, recent memory impairment, or clinically significant head injury.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Adverse event monitoring | From Baseline up to 20 days
Assessment of vital signs (blood pressure, pulse and body temperature) and physical exams | From Baseline up to 20 days
Clinical laboratory tests (chemistry, hematology, urinalysis, renal safety) | From Baseline up to 20 days
Assessment of 12-lead digital electrocardiograms to measure rhythm, rate, morphology, QT/QTc interval | Fron Baseline up to 20 days
Assessment of telemetry, as reported by Investigator Columbia-Suicide Severity Rating Scale (C-SSRS) | From Baseline up to 20 days
  Columbia-Suicide Severity Rating Scale (C-SSRS) captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. Some questions are yes/no and some are on a scale of 1 (low severity) to 5 (high severity). Completed suicide and non-fatal suicide events are yes/no questions and results presented are the number of participants with these events. Worsening of suicidal ideation was an increase in severity of suicidal ideation from baseline.

SECONDARY OUTCOMES:
Investigation of the effect of AZD3293 on plasma and cerebrospinal fluid (CSF) biomarkers relevant for Alzheimer Disease (AD) | Up to 17 days
Investigation of the effect of AZD3293 on plasma and cerebrospinal fluid (CSF) biomarkers relevant for Alzheimer Disease (AD) in mild-moderate AD patients in comparison to elderly healthy volunteers | Up to 17 days
Investigation of the multiple dose Pharmacokinetics for AZD3293 and its metabolite AZ13569724, including dose proportionality for AZD3293 following oral administration | Up 17 days
Investigation of the Pharmacokinetics/Pharmacodynamics relationship of the effect of AZD3293 on biomarkers relevant for Alzheimer Disease (AD) in plasma | Up to 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Alexander, MD, Study Director — AstraZeneca; David Han, MD, Principal Investigator — PAREXEL/CCT Early Phase Clinical Unit
Locations (1):
- Research Site, Glendale, California, United States

REFERENCES:
- [Derived] Cebers G, Lejeune T, Attalla B, Soderberg M, Alexander RC, Budd Haeberlein S, Kugler AR, Ingersoll EW, Platz S, Scott CW. Reversible and Species-Specific Depigmentation Effects of AZD3293, a BACE Inhibitor for the Treatment of Alzheimer's Disease, Are Related to BACE2 Inhibition and Confined to Epidermis and Hair. J Prev Alzheimers Dis. 2016;3(4):202-218. doi: 10.14283/jpad.2016.119. PMID 29199322